CLINICAL TRIAL: NCT00189059
Title: Effects of Pain and the Treatment of Pain With Amitriptyline on Driving Performance, Attentional Capacity and Psychomotor Performance in Chronic Neuropathic Pain Patients
Brief Title: Effects of Amitriptyline for the Treatment of Pain on Driving Performance and Cognition.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Utrecht University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01/341-E
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-04

CONDITIONS: Chronic Neuropathic Pain
Keywords: neuropathic pain; erp; driving; attention; amitriptyline
MeSH Terms: conditions — Neuralgia | interventions — Amitriptyline

INTERVENTIONS:
Drug: amitriptyline

SUMMARY:
The acute and subchronic effects of amitriptyline were compared to placebo in a double-blind crossover randomized study on driving ability and driving-related skills in chronic neuropathic pain patients.It was hypothesized that nocturnally administered 25 mg amitriptyline might affect driving performance negatively after acute, but not after subchronic treatment.

DETAILED DESCRIPTION:
The present study was designed to determine the effects of nocturnally administered 25 mg amitriptyline, compared to placebo, after single (Day 1, acute effects) and repeated (Day 15, subchronic effects) administration on driving performance in neuropathic pain patients. In addition to the on-the-road driving test, laboratory tests measuring driving-related skills were administered. Moreover, effects of amitriptlyine on an attentional capacity task were tested using Event-Related Potentials (ERPs). It was hypothesized that nocturnally administered 25 mg amitriptyline might affect driving performance negatively after acute, but not after subchronic treatment.

ELIGIBILITY:
Inclusion Criteria:

* age, amitriptyline responder, adequately treated with amitriptyline in studied dose before study participation, pain intensity score (VAS) of at least 4 cm on a 10 cm scale, driving licence, driving experience, speak fluently Dutch, normal vision, right-handed

Exclusion Criteria:

* psychological or physical disorder other than pain(-related), other psychotropic medication use, excessive drinking or smoking, alcohol- or drug dependence, illigal drug use

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2002-10; Study Completion 2005-05

PRIMARY OUTCOMES:
driving parameters

SECONDARY OUTCOMES:
laboratory task parameters
ERPs

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Volkerts, PhD, Principal Investigator — University of Utrecht, department of Psychopharmacology
Locations (1):
- University of Utrecht, Utrecht, Utrecht, Netherlands